CLINICAL TRIAL: NCT04170946
Title: A Phase I Study of Talazoparib and Consolidative Thoracic Radiotherapy for Extensive Stage Small Cell Lung Cancer
Brief Title: Talazoparib and Thoracic RT for ES-SCLC
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UHN REB 19-5621
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Lung Cancer; Small-Cell Lung Cancer
Keywords: Talazoparib; Thoracic Radiotherapy; Chemotherapy
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma | interventions — talazoparib; Radiotherapy

STUDY DESIGN:
Intervention Model Description: Dose escalation based on the maximum tolerated dose from each previous cohort within the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Talazoparib in Combination with Low Dose RT (Experimental): Patients will start on talazoparib on day 1 of study intervention, and will continue to orally take talazoparib until the last day of RT (until day 20-23). Patient will start low dose RT on day 6-9, and will continue for 10 fractions throughout 2 weeks. Talazoparib dose levels will start at 0.5mg daily and increase to 1mg if dose limiting toxicites are not observed. Toxicities include renal impairment and other treatment related toxicities Grade ≥3. Patients will be monitored weekly during study treatment, and followed up at 3 weeks, and every 3 months after for 1 year.
  Interventions: Other: Talazoparib in Combination with Low Dose Radiotherapy (RT)

INTERVENTIONS:
Other: Talazoparib in Combination with Low Dose Radiotherapy (RT) — Dose escalation model to determine the safety and MTD of talazoparib in combination with low dose RT.

SUMMARY:
This is a phase I, dose escalating study evaluating the safety of combining talazoparib and low dose consolidative thoracic radiotherapy for small cell lung cancer patients. This study will also determine the maximum tolerated dose (MTD) of talazoparib in combination with low dose thoracic radiotherapy.

Patients will start on talazoparib on day 1 of study intervention, and will continue to orally take talazoparib until the last day of radiation therapy. Up to 24 patients will be enrolled to the study, where the first 3 patients will start with a starting dose level of talazoparib is 0.5 mg PO once daily. This will increase to 1mg daily with each new cohort.

DETAILED DESCRIPTION:
This is a phase I, dose escalating study evaluating the safety of combination talazoparib and low dose consolidative thoracic radiotherapy for extensive-stage small cell lung cancer patients with at least stable disease after standard of care 4 - 6 cycles of chemotherapy (a platinum agent and etoposide). This study will also determine the maximum tolerated dose (MTD) of talazoparib in combination with low dose thoracic radiotherapy. Secondary objectives will be to examine clinical outcomes, including locoregional recurrence within the radiation field, progression-free survival, overall survival and acute/chronic toxicities up to 1 year.

Patients will start on talazoparib on day 1 of study intervention, and will continue to orally take talazoparib until the last day of RT. Patient will start low dose RT on day 6-9, and will continue for 10 fractions throughout 2 weeks. Up to 24 patients will be enrolled to the study, where the first 3 patients will start with a starting dose level of talazoparib is 0.5 mg PO once daily. This will increase to 1mg daily with each new cohort. Patients will be monitored weekly during study treatment, and followed up at 3 weeks, and every 3 months after for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histological documented diagnosis of SCLC confirmed by a UHN pathologist.
* Documented extensive disease
* Completion of induction chemotherapy, 4-6 cycles of a platinum agent and etoposide.
* No disease progression (i.e.SD or better response by RECIST 1.1) at the completion of chemotherapy.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2 (Karnosfsky Performance Score (KPS) ≥50; see Appendix B).
* Adequate organ and marrow function,
* Postmenopausal or evidence of non-childbearing status for women of childbearing potential negative urine or serum pregnancy test within 28 days of study treatment and confirmed prior to treatment on day 1.

Exclusion Criteria:

* Untreated brain metastases.
* Previous radiotherapy to thorax (prior breast RT is permitted).
* Patients receiving any systemic chemotherapy, radiotherapy or immunotherapy (except for standard of care treatments or palliative reasons) within 3 weeks prior to study treatment.
* Exposure to an investigational product within 30 days or 5 half-lives (whichever is longer) prior to start of the current study drug.
* Any previous treatment with PARP inhibitor, including talazoparib.
* Concomitant use of strong P-gp inhibitors
* Concomitant use of other known P-gp inhibitors, P-gp inducers, or BCRP inhibitors
* Persistent toxicities (>Common Terminology Criteria for Adverse Event (CTCAE) grade 2) caused by previous cancer therapy, excluding alopecia.
* Patients with myelodysplastic syndrome/acute leukaemia or with features suggestive thereof.
* Major surgery within 2 weeks of study treatment initiation and patients must have recovered from any effects of any major surgery.
* Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active/uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on High Resolution Computed Tomography (HRCT) scan or any psychiatric disorder that prohibits obtaining informed consent
* Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
* Immunocompromised patients,
* Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT).
* Whole blood transfusions in the last 120 days prior to entry to the study
* Other malignancy within the last 5 years
* Patients with spinal cord compression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-10-05 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Safety of Talazoparib in Combination with Low Dose Thoracic Radiotherapy | Up to 3 years upon enrollment
  Safety will be measured by assessing all adverse events as determined by the investigator using CTCAE v.5.0.
Maximum Tolerated Dose (MTD) of Talazoparib in Combination with Low Dose Thoracic Radiotherapy | Up to 1 year
  MTD will be defined as the maximum dose by a standard 3+3 design

SECONDARY OUTCOMES:
Loco-regional Recurrence | 6 months and 1 year
  Loco-regional recurrence will be assessed by using RECIST v1.1 criteria
Progression-Free Survival (PFS) | 6 months and 1 year
  PFS will be defined as the time of start of radiotherapy to first local/loco-regional or distance recurrence event, or death.
Overall Survival (OS) | 6 months and 1 year
  OS will be defined as the time from the start of radiotherapy to death from any cause.
Acute Toxicities | Up to 1 year
  Acute toxicities will be assessed by physician-graded CTCAE.
Chronic Toxicities | Up to 1 year
  Chronic toxicities will be assessed by physician-graded CTCAE.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Lok, MD, Principal Investigator — Princess Margaret Cancer Center
Locations (1):
- Princess Margaret Cancer Center, University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No